CLINICAL TRIAL: NCT01192932
Title: Effects of Nycthemeral Variations on CT Parameters Reflecting Airways Remodelling, and Pulmonary Emphysema Extent in COPD: Comparisons Between CT Scans Obtained in the Morning and in the Afternoon and Relationships With Pulmonary Function Tests
Brief Title: Effects of Nycthemeral Variations on Computed Tomography (CT) Parameters Reflecting Airways Remodelling, and Pulmonary Emphysema Extent in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Collaborators: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Maxime HACKX, Maxime HACKX, MD, Erasme University Hospital
Other Study IDs: AK/10-02-13/3863
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: COPD; CT; Nycthemeron
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD: COPD patients aged 40 or more, with a smoking history of > 10 pack-years, a post-bronchodilator FEV1/VC < 0.7 and an optimal treatment according to GOLD guidelines will be included. Exclusion criteria are: COPD exacerbation or respiratory infection in the 4 weeks before the begin of the study, concomitant pulmonary disease (tuberculosis, significant bronchiectasis, lung cancer), pulmonary resection, active malignancy or malignancy of any organ system within the past 5 years.
  Interventions: Radiation: Chest CT scan

INTERVENTIONS:
Radiation: Chest CT scan — Supine CT scan after full inspiration. Acquisition parameters: (Topogram 35 mA 120 kV 512 mm length)
  * 90 quality ref mAs with care-dose ON
  * 120 kV
  * Pitch 1.4
  * Rotation time 0.33 s
  * Acquired images 64 x 0.6 mm

SUMMARY:
Computed tomography (CT) studies considering bronchial dimensions in chronic obstructive pulmonary disease (COPD) have never considered nycthemeral variations. Airway calibre, in COPD patients, exhibits a nycthemeral variations with maximal values around noon and minimal values in the early morning, that persists under long-acting bronchodilator. Furthermore, no study has assessed the possible nycthemeral variations of CT scans parameters reflecting airway remodelling and emphysema extent in COPD patients.

This is a prospective study whose purpose is to assess these variations and their relationships with pulmonary function testing (PFT) in COPD patients.

DETAILED DESCRIPTION:
Patients : COPD patients aged 40 years or more, with a smoking history of > 10 pack-years (PY), a post-bronchodilator forced expiratory volume in one second to vital capacity ratio (FEV1/VC) < 0.7 and an optimal treatment according to GOLD guidelines will be included. Exclusion criteria are: COPD exacerbation or respiratory infection in the 4 weeks before the begin of the study, concomitant pulmonary disease (tuberculosis, significant bronchiectasis, lung cancer), pulmonary resection, active malignancy or malignancy of any organ system within the past 5 years.

Procedures: All measurements will be performed on the same day, after obtaining the written informed consent of the patient. Medical history, smoking status and patient's treatment will be collected.

At 08:00 AM (T0): PFT will be performed, including vital capacity (VC), forced vital capacity (FVC), functional residual capacity (FRC), total lung capacity (TLC), residual volume (RV), forced expiratory volume in one second (FEV1), diffusion lung capacity for carbon monoxide (DLCO), and alveolar volume (VA) measurements (either in absolute values and percentage of predicted values). A first CT scan will be performed using the following technique:

* Supine CT scan after full inspiration.
* Acquisition parameters: (Topogram 35 mA 120 kV 512 mm length) 90 quality ref mAs with care-dose ON 120 kV Pitch 1.4 Rotation time 0.33 s Acquired images 64 x 0.6 mm
* Reconstructions parameters: B60f 1mm-thick every 0.7 mm, B20f 1mm-thick every 10.0 mm, B35f 1mm-thick every 0.7 mm, B60f 5mm-thick every 5.0 mm and B35f 5mm-thick every 5.0 mm

At 04:00 PM (T0+8h): PFT will be performed, including vital capacity (VC), forced vital capacity (FVC), functional residual capacity (FRC), total lung capacity (TLC), residual volume (RV), forced expiratory volume in one second (FEV1), diffusion lung capacity for carbon monoxide (DLCO), and alveolar volume (VA) measurements (either in absolute values and percentage of predicted values). A second CT scan will be performed using the following technique:

* Supine CT scan after full inspiration.
* Acquisition parameters: (Topogram 35 mA 120 kV 512 mm length) 90 quality ref mAs with care-dose ON 120 kV Pitch 1.4 Rotation time 0.33 s Acquired images 64 x 0.6 mm
* Reconstructions parameters: B60f 1mm-thick every 0.7 mm, B20f 1mm-thick every 10.0 mm, B35f 1mm-thick every 0.7 mm, B60f 5mm-thick every 5.0 mm and B35f 5mm-thick every 5.0 mm

Data analysis:

* Emphysema index: from B20f reconstructions, calculation of RA960 using Pulmo CT software.
* Airway index: from B60f reconstructions (1mm-thick every 0.7 mm), calculations of luminal area and wall area for several bronchi.

Statistical analyses : Comparisons of CT parameters values or derived values (for example : wall area to airway area ratio) reflecting emphysema and airways remodelling measured on CT scans obtained à T0 and T0+8h. Correlations with PFT values and derived values.

ELIGIBILITY:
Inclusion Criteria:

* age 40 or more
* smoking history > 10 pack-years
* post bronchodilator FEV1/VC < 0.7
* optimal treatment according to GOLD guidelines

Exclusion Criteria:

* COPD exacerbation or infection in the 4 weeks before the study
* concomitant pulmonary disease (tuberculosis, significant bronchiectasis, lung cancer)
* pulmonary resection
* active malignancy or malignancy of any organ system within the past 5 years

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients aged 40 or more, with a smoking history of > 10 PY, a post-bronchodilator FEV1/VC < 0.7 and an optimal treatment according to GOLD guidelines will be included. Exclusion criteria are: COPD exacerbation or respiratory infection in the 4 weeks before the begin of the study, concomitant pulmonary disease (tuberculosis, significant bronchiectasis, lung cancer), pulmonary resection, active malignancy or malignancy of any organ system within the past 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Results of CT Thorax parameters reflecting emphysema and airway remodelling | 4 hours
  Data analysis:
  * Emphysema index: from B20f reconstructions, calculation of RA960 using Pulmo CT software.
  * Airway index: from B60f reconstructions (1mm-thick every 0.7 mm), calculations of luminal area and wall area for several bronchi.

SECONDARY OUTCOMES:
Results of pulmonary function tests | 4 hours
  Pulmonary function tests will be performed in the morning (T0) and in the afternoon (T0+8h): vital capacity (VC), forced vital capacity (FVC), functional residual capacity (FRC), total lung capacity (TLC), residual volume (RV), forced expiratory volume in one second (FEV1), diffusion lung capacity for carbon monoxide will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Alain GEVENOIS, MD, PhD, Study Director — Erasme University Hospital
Locations (1):
- C.H.U Saint-Pierre, Brussels, Belgium

REFERENCES:
- [Background] Nakano Y, Muro S, Sakai H, Hirai T, Chin K, Tsukino M, Nishimura K, Itoh H, Pare PD, Hogg JC, Mishima M. Computed tomographic measurements of airway dimensions and emphysema in smokers. Correlation with lung function. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1102-8. doi: 10.1164/ajrccm.162.3.9907120. PMID 10988137
- [Background] Hasegawa M, Nasuhara Y, Onodera Y, Makita H, Nagai K, Fuke S, Ito Y, Betsuyaku T, Nishimura M. Airflow limitation and airway dimensions in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2006 Jun 15;173(12):1309-15. doi: 10.1164/rccm.200601-037OC. Epub 2006 Mar 23. PMID 16556695
- [Background] Patel BD, Coxson HO, Pillai SG, Agusti AG, Calverley PM, Donner CF, Make BJ, Muller NL, Rennard SI, Vestbo J, Wouters EF, Hiorns MP, Nakano Y, Camp PG, Nasute Fauerbach PV, Screaton NJ, Campbell EJ, Anderson WH, Pare PD, Levy RD, Lake SL, Silverman EK, Lomas DA; International COPD Genetics Network. Airway wall thickening and emphysema show independent familial aggregation in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Sep 1;178(5):500-5. doi: 10.1164/rccm.200801-059OC. Epub 2008 Jun 19. PMID 18565956
- [Background] Berger P, Perot V, Desbarats P, Tunon-de-Lara JM, Marthan R, Laurent F. Airway wall thickness in cigarette smokers: quantitative thin-section CT assessment. Radiology. 2005 Jun;235(3):1055-64. doi: 10.1148/radiol.2353040121. Epub 2005 Apr 15. PMID 15833982
- [Background] Orlandi I, Moroni C, Camiciottoli G, Bartolucci M, Pistolesi M, Villari N, Mascalchi M. Chronic obstructive pulmonary disease: thin-section CT measurement of airway wall thickness and lung attenuation. Radiology. 2005 Feb;234(2):604-10. doi: 10.1148/radiol.2342040013. PMID 15671010
- [Background] Postma DS, Koeter GH, vd Mark TW, Reig RP, Sluiter HJ. The effects of oral slow-release terbutaline on the circadian variation in spirometry and arterial blood gas levels in patients with chronic airflow obstruction. Chest. 1985 May;87(5):653-7. doi: 10.1378/chest.87.5.653. PMID 3987377
- [Background] Calverley PM, Lee A, Towse L, van Noord J, Witek TJ, Kelsen S. Effect of tiotropium bromide on circadian variation in airflow limitation in chronic obstructive pulmonary disease. Thorax. 2003 Oct;58(10):855-60. doi: 10.1136/thorax.58.10.855. PMID 14514937